CLINICAL TRIAL: NCT02155465
Title: A Phase 1/2 Trial of Ruxolitinib and Erlotinib in Patients With EGFR-mutant Lung Adenocarcinoma With Acquired Resistance to Erlotinib
Brief Title: Trial of Ruxolitinib and Erlotinib in Patients With EGFR-mutant Lung Adenocarcinoma With Acquired Resistance to Erlotinib
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-043
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2017-10

CONDITIONS: Lung Cancer
Keywords: Ruxolitinib; Erlotinib; EGFR-mutant; 14-043
MeSH Terms: conditions — Lung Neoplasms | interventions — ruxolitinib; Erlotinib Hydrochloride

ARMS (1):
- Ruxolitinib and Erlotinib (Experimental): Phase I The study will follow a standard 3+3 dose escalation trial design. Three to six patients will need to be enrolled at each dose level and assessed for DLT for 1 full cycle (21 days) before a dose escalation decision is made.
  Phase II Once the MTD has been determined, patients will be enrolled in the phase 2 portion of the single-arm, two-stage, open-label study to determine efficacy of erlotinib and ruxolitinib. Patients will receive erlotinib and ruxolitinib at the MTD established in the phase I portion. The patient take their previous dose of erlotinib if it is less than 150mg daily.
  Interventions: Drug: Ruxolitinib; Drug: Erlotinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib 10mg PO BID
  Ruxolitinib 15mg PO BID
  Ruxolitinib 20mg PO BID
Drug: Erlotinib — Erlotinib 150mg PO QD

SUMMARY:
This is a phase 2 study. The goal of this study is to find out what effects, good and/or bad, taking erlotinib and ruxolitinib has on the patients and on lung cancer. Erlotinib and ruxolitinib are FDA approved for other indications, but the use of erlotinib and ruxolitinib together has not been studied before and is not FDA-approved.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic evidence of advanced (non-operable or metastatic) biopsy-proven stage IV or recurrent lung cancer reviewed at MSKCC.
* a documented somatic activating mutation in EGFR (including but not limited to Exon 19 deletion or L858R)
* Radiographic progression during treatment with erlotinib. Prior chemotherapy regimens are permitted.
* Received erlotinib or other EGFR TK treatment for at least 2 weeks prior to enrollment
* Measurable (RECIST 1.1) indicator lesion not previously irradiated
* Must have undergone biopsy after development of acquired resistance to erlotinib (which is performed as standard of care) with adequate tissue to determine EGFR T790M and tumor histology. Slides from an outside institution may be used.
* KPS ≥ 70%
* Age>18 years old
* Patients must have adequate organ function:

  * AST, ALT, Alk phos ≤ 3.0 x ULN
  * Total bilirubin ≤ 2.0 x ULN
  * Creatinine <2.0 X upper limit of normal and/or a creatinine clearance ≥ 60ml/min
  * Absolute neutrophil count (ANC) ≥1,000 cells/mm³.
  * Platelet count ≥ 100,000/mm³
  * Hemoglobin ≥ 9.0g/dL.

Exclusion Criteria:

* Concurrent therapy with a potent CYP3A4 inducer or inhibitor. Subjects may enter screening when therapy with the potent inhibitor or inducer is completed and may begin study treatment after 1 week or 5 half-lives, whichever is longer.
* Patients with symptomatic brain metastasis requiring escalating doses of steroids.
* Any type of systemic therapy (chemotherapy or experimental drugs) within 3 weeks of starting treatment on protocol except for erlotinib or other EGFR TKI.
* Any radiation within 2 weeks prior to starting treatment on protocol
* Patients with ≥ grade 2 or greater diarrhea despite maximal medical management due to medications or a medical condition such as Crohn's disease, malabsorption.
* Inadequate recovery from any toxicities related to prior treatment (to Grade 1 or baseline).
* Pregnant or lactating women
* Patients who have received prior treatment with JAK inhibitor
* Previously or current malignancies at other sites within the last 2 years, with the exception of adequately treated in situ carcinoma of the cervix, basal or squamous cell carcinoma of the skin, prostate cancer that does not require active treatment per National Comprehensive Cancer Network (NCCN) guidelines, superficial bladder cancer or other noninvasive indolent or stage 1 malignancy without sponsor approval.
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months from Day 1 of study drug administration, New York Heart Association Class III or IV congestive heart failure, or symptomatic arrythmias requiring therapy,
* Chronic or current active infections requiring systemic antibiotics, antifungals or antiviral therapy.
* Known human immunodeficiency virus infection, or hepatitis B virus (HBV) viremia or hepatitis C virus (HCV) viremia. Screening for the study does not require assessment for these infections if not already known.
* Any other condition that, in the opinion of the Investigator, may compromise the safety, compliance of the patient, or would preclude the patient from successful completion of the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Level 1: Level 1 (10mg Ruxolitinib PO bid/ 150mg PO qd Erlotinib)
- Phase 1: Level 2: Level 2 (15mg Ruxolitinib PO bid/ 150mg PO qd Erlotinib)
- Phase 1: Level 3: Level 3 (20mg Ruxolitinib PO bid/ 150mg PO qd Erlotinib)
- PHASE 2: 20mg Ruxolitinib PO BID/ 75 mg Erlotinib PO QD: 20mg Ruxolitinib PO BID/ 75 mg Erlotinib PO QD
- PHASE 2: 20mg Ruxolitinib PO BID / 50 mg Erlotinib PO qd: 20mg Ruxolitinib PO BID / 50 mg Erlotinib PO qd
- PHASE 2 MTD: 20mg Ruxolitinib PO BID / 150 mg Erlotinib PO qd: 20mg Ruxolitinib PO BID / 150 mg Erlotinib PO qd
- PHASE 2 MTD: 20mg Ruxolitinib PO BID / 100 mg Erlotinib PO qd: 20mg Ruxolitinib PO BID / 100 mg Erlotinib PO qd
Period: Overall Study
Arm/Group | Phase 1: Level 1 | Phase 1: Level 2 | Phase 1: Level 3 | PHASE 2: 20mg Ruxolitinib PO BID/ 75 mg Erlotinib PO QD | PHASE 2: 20mg Ruxolitinib PO BID / 50 mg Erlotinib PO qd | PHASE 2 MTD: 20mg Ruxolitinib PO BID / 150 mg Erlotinib PO qd | PHASE 2 MTD: 20mg Ruxolitinib PO BID / 100 mg Erlotinib PO qd
Started | 3 | 3 | 6 | 2 | 1 | 2 | 5
Completed | 3 | 3 | 6 | 2 | 1 | 2 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Level 1 | Phase 1: Level 2 | Phase 1: Level 3 | Phase 2: 20mg Ruxolitinib PO BID/ 75 mg Erlotinib PO QD | PHASE 2: 20mg Ruxolitinib PO BID / 50 mg Erlotinib PO qd | PHASE 2 MTD: 20mg Ruxolitinib PO BID / 150 mg Erlotinib PO qd | PHASE 2 MTD: 20mg Ruxolitinib PO BID / 100 mg Erlotinib PO qd | Total
Number analyzed (Participants) | 3 | 3 | 6 | 2 | 1 | 2 | 5 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 5 | 1 | 0 | 0 | 3 | 12
  >=65 years | 1 | 2 | 1 | 1 | 1 | 2 | 2 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 1 | 1 | 0 | 4 | 13
  Male | 1 | 2 | 2 | 1 | 0 | 2 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  White | 2 | 2 | 5 | 1 | 1 | 2 | 4 | 17
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6 | 2 | 1 | 2 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Maximally Tolerated Dose (MTD) (Phase I)
Time Frame: 1 year
Population: Maximally Tolerated Dose (MTD) is determined by evaluating all Phase I participants as a whole. All Phase I participants are evaluated together to determine the MTD.
Measure: Number; unit: mg
Groups:
- Phase I Participants: Phase I The study will follow a standard 3+3 dose escalation trial design. Three to six patients will need to be enrolled at each dose level and assessed for DLT for 1 full cycle (21 days) before a dose escalation decision is made.
- Phase II Participants: Phase II Once the MTD has been determined, patients will be enrolled in the phase 2 portion of the single-arm, two-stage, open-label study to determine efficacy of erlotinib and ruxolitinib. Patients will receive erlotinib and ruxolitinib at the MTD established in the phase I portion. The patient take their previous dose of erlotinib if it is less than 150mg daily.
Arm/Group | Phase I Participants | Phase II Participants
Number analyzed (Participants) | 12 | 0
mg
  Erlotinib Daily | 150 |
  Ruxolitinib Twice Daily | 20 |

2. Primary Outcome: Assess Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions; Progressive disease (PD), at least a 20% increase in the sum of the diameter of the target lesions or the appearance of one or more new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD
Time Frame: 1 year
Population: Participants response to study treatment were combined and evaluated to determine an overall response rate.
Measure: Number (95% Confidence Interval); unit: % of participants with partial response
Arm/Group | Ruxolitinib and Erlotinib
Number analyzed (Participants) | 22
% of participants with partial response | 5 [0 to 13]

3. Secondary Outcome: Number of Participants With NCI CTCAE Toxicity
Description: Toxicity grading will be performed in accordance with NCI CTCAE, version 4.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Level 1: 10mg Ruxolitinib PO bid/ 150mg PO qd Erlotinib
- Phase 1: Level 2: 15mg Ruxolitinib PO bid/ 150mg PO qd Erlotinib
- Phase 1: Level 3: 20mg Ruxolitinib PO bid/ 150mg PO qd Erlotinib
Arm/Group | Phase 1: Level 1 | Phase 1: Level 2 | Phase 1: Level 3 | Phase 2: 20mg Ruxolitinib PO BID/ 75 mg Erlotinib PO QD | Phase 2: 20mg Ruxolitinib PO BID / 50 mg Erlotinib PO qd | PHASE 2 MTD: 20mg Ruxolitinib PO BID / 150 mg Erlotinib PO qd | PHASE 2 MTD: 20mg Ruxolitinib PO BID / 100 mg Erlotinib PO qd
Number analyzed (Participants) | 3 | 3 | 6 | 2 | 1 | 2 | 5
Participants | 3 | 3 | 6 | 2 | 1 | 2 | 5

4. Secondary Outcome: Progression-free Survival
Time Frame: 2 years
Population: Participants response to study treatment were combined and evaluated to determine an overall progression-free survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ruxolitinib and Erlotinib
Number analyzed (Participants) | 22
months | 2.2 [1.5 to 4.1]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Phase 1: Level 1 | Phase 1: Level 2 | Phase 1: Level 3 | PHASE 2: 20mg Ruxolitinib PO BID/ 75 mg Erlotinib PO QD | PHASE 2: 20mg Ruxolitinib PO BID / 50 mg Erlotinib PO qd | PHASE 2 MTD: 20mg Ruxolitinib PO BID / 150 mg Erlotinib PO qd | PHASE 2 MTD: 20mg Ruxolitinib PO BID / 100 mg Erlotinib PO qd
All-Cause Mortality (participants affected / at risk) | 3/3 | 1/3 | 5/6 | 2/2 | 1/1 | 1/2 | 3/5
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 2/6 | 0/2 | 1/1 | 0/2 | 1/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 5/6 | 2/2 | 1/1 | 2/2 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Level 1 (N=3) | Phase 1: Level 2 (N=3) | Phase 1: Level 3 (N=6) | PHASE 2: 20mg Ruxolitinib PO BID/ 75 mg Erlotinib PO QD (N=2) | PHASE 2: 20mg Ruxolitinib PO BID / 50 mg Erlotinib PO qd (N=1) | PHASE 2 MTD: 20mg Ruxolitinib PO BID / 150 mg Erlotinib PO qd (N=2) | PHASE 2 MTD: 20mg Ruxolitinib PO BID / 100 mg Erlotinib PO qd (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | NA | 0 | NA | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | NA | 0 | NA | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | NA | 0 | NA | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | 0 | NA | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | NA | 0 | NA | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | NA | 0 | NA | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | NA | 1 | NA | 0
Fatigue (General disorders) | 1 | 0 | 0 | NA | 0 | NA | 0
Fever (General disorders) | 0 | 0 | 1 | NA | 0 | NA | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | NA | 0 | NA | 1
Neoplasms ben/mal/unk (inc cyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | NA | 0 | NA | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | NA | 1 | NA | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | NA | 0 | NA | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | 1 | NA | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | 0 | NA | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | NA | 0 | NA | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | NA | 0 | NA | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Level 1 (N=3) | Phase 1: Level 2 (N=3) | Phase 1: Level 3 (N=6) | PHASE 2: 20mg Ruxolitinib PO BID/ 75 mg Erlotinib PO QD (N=2) | PHASE 2: 20mg Ruxolitinib PO BID / 50 mg Erlotinib PO qd (N=1) | PHASE 2 MTD: 20mg Ruxolitinib PO BID / 150 mg Erlotinib PO qd (N=2) | PHASE 2 MTD: 20mg Ruxolitinib PO BID / 100 mg Erlotinib PO qd (N=5)
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 2 | 1 | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell decreased (Investigations) | 0 | 0 | 2 | 1 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 2 | 0 | 1 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 3 | 0 | 1 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 3 | 1 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
INR increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localized edema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT02155465/Prot_SAP_000.pdf